CLINICAL TRIAL: NCT06165341
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Safety and Efficacy of Fazirsiran in the Treatment of Alpha-1 Antitrypsin Deficiency-Associated Liver Disease With METAVIR Stage F1 Fibrosis
Brief Title: Study to Learn About the Safety of Fazirsiran and if it Can Help People With Alpha-1 Antitrypsin Liver Disease With Mild Liver Scarring (Fibrosis)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-999-3002; 2023-504198-19-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Alpha1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fazirsiran 200 mg (Experimental): Participants will receive fazirsiran 200 milligrams (mg), injection, subcutaneously on Day 1, at Week 4 and then every 12 weeks (Q12W) for up to Week 100.
  Interventions: Drug: Fazirsiran Injection
- Placebo (Placebo Comparator): Participants will receive fazirsiran matching placebo injection, subcutaneously on Day 1, at Week 4 and Q12W for up to Week 100.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fazirsiran Injection — Fazirsiran will be injected subcutaneously.
  Other Names: TAK-999; ARO-AAT; ADS-001
  Arms: Fazirsiran 200 mg
Drug: Placebo — Fazirsiran matching placebo.
  Arms: Placebo

SUMMARY:
The liver produces a protein called alpha-1 antitrypsin (AAT). AAT is normally released into the bloodstream. In some people, the liver makes an abnormal version of the AAT protein, called Z-AAT. Making an abnormal version of the AAT protein can result in liver disease as Z-AAT builds up in liver cells, which leads to liver problems such as liver scarring (fibrosis), continuing liver damage (cirrhosis), and eventually end stage liver disease. Fazirsiran is a medicine that reduces the creation of the Z-AAT protein and thus the build-up of this abnormal protein in the liver. People with this type of liver disease who already have mild liver scarring will take part in the study. They will be treated with fazirsiran or a placebo for about 2 years. This study will check the long-term safety of fazirsiran, whether participants tolerate the treatment and if there are any effects on liver scarring. A liver biopsy, a way of collecting a small tissue sample from the liver, will be taken twice during the study.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, the participant is capable of understanding and fully complying with the protocol requirements and adhering to the protocol schedule.
* The participant is able to read, understand, and complete the study questionnaires electronically per the investigator's judgment.
* The participant signs and dates a written Informed Consent Form (ICF). Any required privacy authorization should also be signed before the initiation of any study procedures.
* The participant, of any sex, is aged 18 to 75 years, inclusive.
* The participant must have a diagnosis of the protease inhibitor Z mutation (PiZZ) genotype AATD. A diagnosis of PiZZ from source-verifiable medical records is permitted. Otherwise, participants must undergo PiZZ confirmatory testing (genotyping for PiS and PiZ alleles) at screening. PiMZ or PiSZ genotypes are not permitted.
* The participant's liver biopsy core samples collected as per protocol requirements.
* The participant has evidence of METAVIR stage F1 liver fibrosis, evaluated by a centrally read baseline liver biopsy during the screening period; or confirmed as meeting all the entry criteria by central reading from a previous biopsy conducted within 1 year before the estimated enrollment date using an adequate liver biopsy and slides as defined in the study laboratory manual.
* The participant has a pulmonary status that meets the protocol requirements.
* It must be confirmed that the participant does not have hepatocellular carcinoma (HCC).
* Any participant who is taking statins, angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, or beta-1 selective adrenergic receptor inhibitors must have been receiving a stable dose of these medications for at least 8 weeks before randomization. All attempts are to be made for the participant to continue the same dose of the medication for the duration of study participation.
* An adult participant must have a body mass index (BMI) between 18 and 39 kilogram per meter square (kg/m^2), inclusive.
* The participant has a 12-lead electrocardiogram at screening that, in the opinion of the investigator, has no abnormalities that could compromise the participant's safety in this study.
* The participant is a nonsmoker.
* If the participant was being treated with any respiratory medications including inhaled bronchodilators, inhaled anticholinergics, inhaled corticosteroids, or low-dose systemic corticosteroids (prednisone less than or equal to [<=10] milligrams per day [mg/d] or its equivalent), the doses of the participant's medications must have remained unchanged for greater than or equal to (>=) 4 weeks before screening.
* The participant must have suitable venous access for blood sampling.
* A person of childbearing potential (POCBP) must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 before dosing.
* The participant must use appropriate contraception methods (that is, highly effective methods for female and medically appropriate methods for male study participants) for the entire duration of the study and for 6 months after the last dose of study medication. The participant must not donate sperm for at least 6 months after the last dose of study medication.

Exclusion criteria:

* The participant has evidence of >= F2 fibrosis based on liver biopsy during the screening period.
* The participant has a history of liver decompensating events.
* The participant has a history of varices based on a previous esophagogastroduodenoscopy.
* The participant has portal vein thrombosis.
* The participant has undergone a prior trans-jugular portosystemic shunt procedure.
* The participant has evidence of other forms of chronic liver diseases.
* The participant has a history of malignancy within the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer. Participants with curatively treated malignancies who have no evidence of metastatic disease and disease-free interval greater than (>) 1 year may be enrolled after approval by the medical monitor.
* The participant has an abnormal finding of clinical relevance at the screening evaluation and before administration of the first dose of study dosing that, in the opinion of the investigator, could adversely impact participant safety during the study or adversely impact study results.
* The participant has any laboratory abnormalities at screening and before the first dose of the study drug that meet protocol parameters.
* The participant is expected to have severe and unavoidable high-level exposure to inhaled pulmonary toxins during the study such as may occur with occupational exposure to mineral dusts or metals.
* The participant has a recent lower respiratory tract infection, such as pneumonia, within the last 6 months before screening. The participant may be screened earlier based on principal investigator (PI) assessment of clinical recovery and return to baseline pulmonary function in discussion with the medical monitor.
* The participant has a history of frequent pulmonary exacerbations (>=2 moderate or severe exacerbations within 52 weeks before screening).
* The participant is experiencing a pulmonary exacerbation at the time of screening (participant may be rescreened after the clinical resolution of an exacerbation).
* The participant is receiving long-term, around-the-clock oxygen supplementation or supplemental oxygen with continuous positive airway pressure (CPAP) or bilevel positive airway pressure for acute respiratory failure. The following conditions are allowable for the participant to enter screening: short-term use of oxygen supplementation (example, for the management of acute chronic obstructive pulmonary disease [COPD] exacerbation) or CPAP for obstructive sleep apnea.
* The participant has human immunodeficiency virus (HIV) infection as shown by the presence of anti-HIV antibody (seropositive).
* The participant is seropositive for hepatitis B virus (HBV surface antigen positive and/or HBV core antibody positive without HBV surface antibody at screening) or hepatitis C virus (HCV) (detectable HCV Ribonucleic Acid [RNA] at screening). Cured HCV (positive antibody test without detectable HCV RNA for at least 6 months after treatment) is acceptable.
* The participant has unstable, poorly controlled, or severe hypertension. Participants may be rescreened once their blood pressure (BP) is successfully controlled.
* The participant has a history of torsades de pointes, ventricular rhythm disturbances (example, ventricular tachycardia), heart block (excluding first-degree block, being PR interval prolongation only), congenital long QT syndrome or new ST-segment elevation or depression or a new Q wave on ECG. Participants with a history of atrial arrhythmias should be discussed with the medical monitor.
* The participant has symptomatic heart failure (per New York Heart Association guidelines), unstable angina, myocardial infarction, severe cardiovascular disease (ejection fraction less than [<] 20 percent [%]), transient ischemic attack, or cerebrovascular accident within 6 months before screening.
* The participant has a history of major surgery within 12 weeks of screening (or longer, at the discretion of the investigator).
* The participant has a history of more than moderate alcohol consumption within 12 months before the screening visit.
* The participant has a history of drug abuse (such as cocaine, phencyclidine) within 1 year before the screening visit or has a positive urine drug screen at screening.
* The participant has previously been treated with fazirsiran or any other RNA interference (RNAi) for alpha-1 antitrypsin deficiency-associated liver disease (AATD-LD).
* The participant has a history of hypersensitivity or allergies with any associated excipients of fazirsiran.
* The participant has received an investigational agent or device within 30 days, or 5 half-lives, whichever is longer, before the dosing of study medication or is currently participating in an investigational study involving a therapeutic intervention.
* The participant has donated >=500 milliliter (mL) of blood within 1 month of the administration of study treatment.
* The participant has any concomitant medical or psychiatric condition or social situation that would make it difficult to comply with protocol requirements or put the participant at additional safety risk. The participant has a history of clinically significant hematologic, renal, hepatic, pulmonary, neurologic, psychiatric, gastrointestinal (GI), systemic inflammatory, metabolic, or endocrine disorder or any other condition that, in the opinion of the investigator, rendered the participant a poor candidate for inclusion into the study.
* The participant has a history of thromboembolic disease (including deep vein thrombosis or pulmonary embolism), within 6 months before screening, or is taking chronic anticoagulants.
* This participant is unable to return for all scheduled study visits.
* The participant has known or suspected coronavirus disease 2019 (COVID-19) that, in the opinion of the sponsor and investigator, does not resolve during screening. Positive antibody testing for COVID-19 without other evidence of current or recent active infection does not exclude participation. Enrollment of participants who fail inclusion due to COVID-19 infection may be temporarily delayed at the discretion of the sponsor and investigator. If the participant has a positive polymerase chain reaction (PCR) with no other evidence of infection, a retest may be allowed; however, to enroll in the study the participant must have a negative PCR.
* The participant is a study site employee involved in the conduct of this study, an immediate family member (example, spouse, parent, child, sibling), is in a dependent relationship with study site employee who is involved in the conduct of this study or may consent under duress.
* The participant takes or is required to take excluded medications.
* The participant is pregnant or breastfeeding or intending to become pregnant before participating in this study, during the study, or within 6 months after last dose of the study drug; or the participant is intending to donate ova during such time period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-08-26 (Estimated); Study Completion 2028-08-26 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | From start of study drug administration up to End of study (EOS) (Week 124)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not it is considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study intervention. An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, suspected transmission of any infectious agent, an important medical event. AEs and SAEs including any pulmonary AEs or SAEs indicative of worsening pulmonary condition (example, pulmonary exacerbation, respiratory infection, significant pulmonary function test decline) will be reported.
Number of Participants With Clinically Significant Change From Baseline in Pulmonary Function Parameters | From start of study drug administration up to EOS (Week 124)
  Standard pulmonary function parameters will be used to study lung function. Clinical significance of pulmonary function parameters will be determined at the investigator's discretion.
Change From Baseline in Whole Lung 15th Percentile Density as Measured by Computed Tomography (CT) Lung Densitometry | Baseline up to Week 100
  Change from baseline in whole lung 15th percentile density as measured by CT lung densitometry will be assessed.
Number of Participants With Clinically Significant Changes in Vital Signs | From start of study drug administration up to EOS (Week 124)
  Vital signs include body temperature, respiratory rate, blood pressure (systolic and diastolic), pulse (beats per minute) and pulse oximetry. Clinical significance of vital signs will be determined at the investigator's discretion.
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Parameters | From start of study drug administration up to EOS (Week 124)
  12-lead ECG will be evaluated. Any clinically significant change in ECG assessments will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters | From start of study drug administration up to EOS (Week 124)
  Laboratory parameters assessments include hematology, biochemistry including liver tests, coagulation, and urinalysis. Clinical significance of laboratory parameters will be determined at the investigator's discretion.

SECONDARY OUTCOMES:
Change From Baseline in Serum Z-AAT Protein Over Time to Week 106 | Baseline up to Week 106
  Change From Baseline in Serum Z-AAT Protein will be assessed.
Percent Change From Baseline in Intrahepatic Liver Z-AAT Protein at Week 106 | Baseline up to Week 106
  Percent change from baseline in intrahepatic liver Z-AAT protein will be assessed.
Change From Baseline in Intrahepatic Z-AAT Protein Polymer Burden Assessed by Periodic Acid Schiff Plus Diastase (PAS+D) Staining in Liver Biopsy at Week 106 | Baseline up to Week 106
  Change from baseline in intrahepatic Z-AAT protein polymer burden assessed by PAS+D staining in liver biopsy will be assessed.
Number of Participants with No Change or Decrease From Baseline in Intrahepatic Z-AAT Protein Polymer Burden Assessed by PAS+D staining at Week 106 | Baseline up to Week 106
  Number of participants with no change or decrease from baseline in intrahepatic Z-AAT protein polymer burden assessed by PAS+D staining will be reported.
Change From Baseline in Intrahepatic Portal Inflammation Score in Liver Biopsy at Week 106 | Baseline up to Week 106
  Change in portal inflammation score in liver biopsy is based on pathology slide reads. Inflammation will be assessed on a scale of 0-3, with higher scores showing more severe inflammation.
Number of Participants with No Change or Decrease From Baseline in Intrahepatic Portal Inflammation Score at Week 106 | Baseline up to Week 106
  No Change or decrease in portal inflammation score is based on pathology slide reads. Inflammation will be assessed on a scale of 0-3, with higher scores showing more severe inflammation. Number of Participants with no change or decrease from baseline in intrahepatic portal inflammation score will be reported.
Number of Participants With No Change or Decrease From Baseline in Histologic Fibrosis Score (Meta-analysis of Histological Data in Viral Hepatitis [METAVIR] Staging ) at Week 106 | Baseline up to Week 106
  No change or decrease in histologic fibrosis (METAVIR staging) will be assessed using a fibrosis score of F0-F4, where higher scores mean a worse result. Number of participants with no change or decrease from baseline in histologic fibrosis score (by [METAVIR] staging) at Week 106 will be reported.
Change From Baseline in Vibration-Controlled Transient Elastography (VCTE)-Derived Liver Stiffness | Baseline up to Week 106
  Change from baseline in VCTE-derived liver stiffness will be assessed.
Change From Baseline in Markers of Liver Injury | Baseline up to Week 106
  Change from baseline in marker (alanine aminotransferase [ALT], aspartate aminotransferase [AST], glutamyl transferase [GGT]) of liver injury will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (20):
  - St Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic - PPDS, Phoenix, Arizona
  - University of Arizona Thomas D. Boyer Liver Institute, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - UCLA Pulmonary and Critical Care, Los Angeles, California
  - University of California Benioff Children's Hospital, San Francisco, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Indiana University School of Medicine-Indianapolis, Indianapolis, Indiana
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Hospital - 1500 E Medical Center Dr, Ann Arbor, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Mayo Clinic PPDS, Rochester, Minnesota
  - NYU Langone Medical Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Texas Liver Institute American Research Corporation, San Antonio, Texas
  - Bon Secours St. Mary's Hospital, Newport, Virginia
- Austria (2):
  - LKH-Universitätsklinikum Graz, Graz
  - KABEG - Klinikum Klagenfurt Am Wörthersee, Klagenfurt
- Belgium (2):
  - UZ Antwerpen, Antwerp
  - UZ Leuven, Leuven
- Inspiration Research Limited, Toronto, Ontario, Canada
- France (3):
  - Hôpital de La Croix Rousse, Lyon
  - Hopital PONTCHAILLOU CHU de Rennes, Rennes
  - Hôpital Paul Brousse, Val-de-Marne
- Germany (4):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Charité - Campus Virchow-Klinikum, Berlin
  - Hannover Medical School, Hanover
  - Universitätsklinikum Tübingen, Tübingen
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- ID Clinic Arkadiusz Pisula, Mysłowice, Poland
- Portugal (3):
  - CCA Hospital Braga, Braga
  - Hospital Dr. Nélio Mendonça, Funchal
  - Centro Hospitalar de Universitário de Santo António E.P.E, Porto
- Hospital Universitario Virgen del Rocio - PPDS, Seville, Spain
- Karolinska Universitetssjukhuset Huddinge, Huddinge, Sweden
- Universitätsspital Bern, Bern, Switzerland
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/4a3e8be16f9a47d2?idFilter=%5B%22TAK-999-3002%22%5D